CLINICAL TRIAL: NCT07236372
Title: Comparative Efficacy of Standard-Dose Versus Updosed Cetirizine in Acute Urticaria: A Randomized Controlled Trial
Brief Title: Comparing Standard-Dose and High-Dose Cetirizine for Acute Urticaria
Acronym: CURE-AU
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Phayao (Other)
Responsible Party: Principal Investigator, Wasuchon Chaichan, Lecturer, Department of Internal Medicine, School of Medicine, University of Phayao, University of Phayao
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HREC-UP-HSST 1.3/002/69; MD68-19 (Other Grant/Funding Number: School of Medicine, University of Phayao)
Record Dates: First submitted 2025-11-15; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Acute Urticaria
Keywords: Acute Urticaria; Updosed Cetirizine; High-Dose Antihistamine; Standard-Dose Cetirizine; Second-Generation Antihistamine; Randomized Controlled Trial
MeSH Terms: interventions — Cetirizine

STUDY DESIGN:
Intervention Model Description: This study uses a randomized, parallel-group design in which participants are assigned in a 1:1 ratio to receive either the standard dose or the high dose of cetirizine. A blinded outcome assessor evaluates symptom improvement to minimize measurement bias. The intervention lasts 7 days, followed by scheduled follow-up visits to assess symptom resolution, recurrence, and safety outcomes.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard-Dose Cetirizine (10 mg/day) (Active Comparator): Participants in this arm will receive standard-dose cetirizine at 10 mg once daily for 7 days. The medication will be provided in capsule form. Participants will record their daily urticaria symptoms and return for scheduled follow-up visits to assess symptom improvement and safety outcomes.
  Interventions: Drug: Cetirizine 10 mg
- Updosed Cetirizine (40 mg/Day) (Experimental): Participants in this arm will receive high-dose cetirizine at 40 mg per day, taken as 20 mg twice daily for 7 days. The medication will be provided in capsule form. Participants will record their daily urticaria symptoms and return for scheduled follow-up visits to assess symptom improvement, the need for rescue medications, and any side effects.
  Interventions: Drug: Cetirizine 40 mg

INTERVENTIONS:
Drug: Cetirizine 10 mg — Participants in the standard-dose arm receive cetirizine 10 mg orally once daily for 7 days. The study medication is provided in capsule form to match the appearance of the high-dose capsules.
  Arms: Standard-Dose Cetirizine (10 mg/day)
Drug: Cetirizine 40 mg — Participants in the high-dose arm receive cetirizine 20 mg orally twice daily (total 40 mg/day) for 7 days. The study medication is provided in capsule form to ensure identical appearance between arms.
  Arms: Updosed Cetirizine (40 mg/Day)

SUMMARY:
The goal of this clinical trial is to learn whether a higher dose of cetirizine works better than the standard dose to relieve symptoms of acute urticaria (hives) in adults. The study also aims to learn about the safety of taking a higher dose for a short period of time.

The main questions the study aims to answer are:

Does the higher dose of cetirizine help people with acute urticaria improve faster than the standard dose? What side effects do participants experience when taking the higher dose?

Researchers will compare two groups:

one group taking the standard dose of cetirizine (10 mg per day) and another group taking a higher dose (40 mg per day). This will help researchers understand which dose works better and whether the higher dose is safe.

Participants will:

Take the assigned study medication for 7 days Record their daily symptoms, including itch and hive severity Return for follow-up visits on Day 3, Day 7, and Week 6 Have blood tests to check liver and kidney function before and after treatment

This study may help improve treatment options for people with acute urticaria and reduce the need for unnecessary steroid use.

DETAILED DESCRIPTION:
This study is a randomized, parallel-group clinical trial designed to evaluate whether a higher dose of cetirizine provides better symptom relief than the standard dose in adults with acute urticaria. Acute urticaria often causes sudden wheals and intense itching that can significantly affect comfort and daily functioning. Although standard-dose second-generation antihistamines are recommended as first-line treatment, many people do not fully improve and are frequently prescribed systemic corticosteroids, which may lead to unnecessary side effects.

This trial investigates whether increasing the dose of cetirizine to 40 mg per day offers faster or more complete symptom improvement without increasing safety risks. Participants will be randomly assigned to receive either the standard dose or the higher dose for 7 days. The study uses a blinded outcome assessment to minimize bias. Symptom severity will be measured using validated tools, and participants will be monitored for side effects throughout the study.

Laboratory tests will be used to assess kidney and liver function before and after treatment. Follow-up visits will evaluate short-term changes in symptoms as well as the potential for recurrence or progression to chronic urticaria. The findings may help guide clinical decision-making and support more rational use of antihistamines while reducing reliance on corticosteroids in acute urticaria care.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 60 years
* Clinical diagnosis of acute urticaria made by a physician
* Onset of new wheals within the past 24 hours
* Able and willing to comply with study procedures, complete symptom diaries, and attend follow-up visits
* Provides written informed consent prior to participation

Exclusion Criteria:

* Use of systemic corticosteroids within the past 5 days
* Use of antihistamines within the past 5 days
* Use of immunosuppressive medications within the past 5 days
* Clinical signs of anaphylaxis, including respiratory distress, hypotension, abdominal pain, or acute laryngeal swelling
* Presence of angioedema without wheals
* Known diagnosis of chronic urticaria
* Known severe renal impairment (creatinine clearance <10 mL/min), heart failure (ejection fraction <40%), or hepatic failure
* Other skin conditions that may interfere with assessment (e.g., atopic dermatitis, eczema, bullous pemphigoid, AGEP)
* Use of ACE inhibitors or ARBs within the past 5 days
* Known allergy or hypersensitivity to cetirizine or components of the study medication
* Pregnancy or breastfeeding
* Known diabetes mellitus
* History of gastrointestinal ulcer disease
* Any condition that, in the investigator's judgment, would interfere with study participation or safety
* Declines to provide informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Time to Resolution of Acute Urticaria Symptoms | From Day 0 (first dose) to Day 7 or until complete symptom resolution, whichever occurs first.
  The time from the first dose of study medication to the complete resolution of acute urticaria symptoms, defined as the absence of hives and an itch score of 0 for at least 24 consecutive hours. Symptom status will be assessed using patient-reported daily symptom diaries and validated scoring tools.
Change in Urticaria Activity Score From Baseline | Baseline to Day 7
  The change in total UAS7 score from baseline to Day 7, based on daily patient-reported wheal and itch scores collected in symptom diaries.

SECONDARY OUTCOMES:
Use of Systemic Corticosteroids as Rescue Medication | Day 0 to Day 7
  The proportion of participants requiring systemic corticosteroids due to persistent or worsening acute urticaria symptoms despite taking the assigned study medication.
Change in Dermatology Life Quality Index (DLQI) | Baseline to Day 7
  The change in Dermatology Life Quality Index (DLQI) from baseline to Day 7 to assess the clinical response and quality of life impact of treatment.
Incidence and Characteristics of Adverse Events | Day 0 to Day 7 and Week 6 follow-up
  Number, type, and severity of adverse events occurring during treatment with standard-dose versus high-dose cetirizine. Adverse events may include sedation, dizziness, or other treatment-related symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Wasuchon Chaichan, Principal Investigator — School of Medicine, University of Phayao
Locations (1):
- University of Phayao Hospital, Phayao, Muang, Thailand

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the dataset contains sensitive health information and the study sample size is small, making de-identification difficult. In addition, the informed consent form does not include permission for public sharing of individual-level data.

REFERENCES:
- [Result] Jamjanya S, Danpanichkul P, Ongsupankul S, Taweesap S, Thavorn K, Hutton B, Ruengorn C, Bernstein JA, Chuamanochan M, Nochaiwong S. Evaluation of Pharmacological Treatments for Acute Urticaria: A Systematic Review and Meta-Analysis. J Allergy Clin Immunol Pract. 2024 May;12(5):1313-1325. doi: 10.1016/j.jaip.2024.01.022. Epub 2024 Jan 25. PMID 38280453
- [Result] Chu X, Wang J, Ologundudu L, Brignardello-Petersen R, Guyatt GH, Oykhman P, Bernstein JA, Saini SS, Beck LA, Waserman S, Moellman J, Khan DA, Ben-Shoshan M, Baker DR, Oliver ET, Sheikh J, Lang D, Mathur SK, Winders T, Eftekhari S, Gardner DD, Runyon L, Asiniwasis RN, Cole EF, Chan J, Wheeler KE, Trayes KP, Tran P, Chu DK. Efficacy and Safety of Systemic Corticosteroids for Urticaria: A Systematic Review and Meta-Analysis of Randomized Clinical Trials. J Allergy Clin Immunol Pract. 2024 Jul;12(7):1879-1889.e8. doi: 10.1016/j.jaip.2024.04.016. Epub 2024 Apr 18. PMID 38642709
- [Result] Badloe FMS, Grosber M, Ring J, Kortekaas Krohn I, Gutermuth J. Treatment of acute urticaria: A systematic review. J Eur Acad Dermatol Venereol. 2024 Nov;38(11):2082-2092. doi: 10.1111/jdv.19904. Epub 2024 Feb 29. PMID 38420865
- [Result] Okubo Y, Shigoka Y, Yamazaki M, Tsuboi R. Double dose of cetirizine hydrochloride is effective for patients with urticaria resistant: a prospective, randomized, non-blinded, comparative clinical study and assessment of quality of life. J Dermatolog Treat. 2013 Apr;24(2):153-60. doi: 10.3109/09546634.2011.608783. Epub 2011 Aug 24. PMID 21810005
- [Result] Zuberbier T, Abdul Latiff AH, Abuzakouk M, Aquilina S, Asero R, Baker D, Ballmer-Weber B, Bangert C, Ben-Shoshan M, Bernstein JA, Bindslev-Jensen C, Brockow K, Brzoza Z, Chong Neto HJ, Church MK, Criado PR, Danilycheva IV, Dressler C, Ensina LF, Fonacier L, Gaskins M, Gaspar K, Gelincik A, Gimenez-Arnau A, Godse K, Goncalo M, Grattan C, Grosber M, Hamelmann E, Hebert J, Hide M, Kaplan A, Kapp A, Kessel A, Kocaturk E, Kulthanan K, Larenas-Linnemann D, Lauerma A, Leslie TA, Magerl M, Makris M, Meshkova RY, Metz M, Micallef D, Mortz CG, Nast A, Oude-Elberink H, Pawankar R, Pigatto PD, Ratti Sisa H, Rojo Gutierrez MI, Saini SS, Schmid-Grendelmeier P, Sekerel BE, Siebenhaar F, Siiskonen H, Soria A, Staubach-Renz P, Stingeni L, Sussman G, Szegedi A, Thomsen SF, Vadasz Z, Vestergaard C, Wedi B, Zhao Z, Maurer M. The international EAACI/GA(2)LEN/EuroGuiDerm/APAAACI guideline for the definition, classification, diagnosis, and management of urticaria. Allergy. 2022 Mar;77(3):734-766. doi: 10.1111/all.15090. Epub 2021 Oct 20. PMID 34536239